CLINICAL TRIAL: NCT06328387
Title: Open, Controlled, Multicenter Phase I/II Clinical Study of Hydroxychloroquine in Combination With Antibody-drug Conjugate Versus Antibody-drug Conjugate for Advanced Breast Cancer.
Brief Title: HCQ+ADC vs ADC in the Treatment of Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jianli Zhao, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-064-03
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Antibody-drug Conjugate; Hydroxychloroquine; Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydroxychloroquine; sacituzumab govitecan; trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: The research model consists of four arms：
  1. arm A: SG.
  2. arm B: HCQ+SG.
  3. arm C: T-DXd .
  4. arm D: HCQ+T-DXd.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sacituzumab Govitecan (Other): Sacituzumab Govitecan (SG) is given by intervenous route, 10 mg/kg on day 1 and day 8 of 21-day treatment cycles. Patient will receive treatment until disease progression, unacceptable toxicity, or decision to withdraw its participation.
  Interventions: Drug: Sacituzumab Govitecan
- Hydroxychloroquine Combined With Sacituzumab Govitecan (Experimental): The dosage of hydroxychloroquine is determined based on the dose escalation study, and the appropriate administration method will be determined based on this result.
  Sacituzumab Govitecan (SG) is given by intervenous route, 10 mg/kg on day 1 and day 8 of 21-day treatment cycles. Patient will receive treatment until disease progression, unacceptable toxicity, or decision to withdraw its participation.
  Interventions: Drug: Hydroxychloroquine; Drug: Sacituzumab Govitecan
- Trastuzumab Deruxtecan (Other): Patients will receive T-DXd at 5.4 mg/kg administered as an intravenous (IV) infusion every three-weeks (Q3W) until disease progression, unacceptable toxicity, death, or discontinuation from the study.
  Interventions: Drug: Trastuzumab Deruxtecan
- Hydroxychloroquine Combined With Trastuzumab Deruxtecan (Experimental): The dosage of hydroxychloroquine is determined based on the dose escalation study, and the appropriate administration method will be determined based on this result.
  Patients will receive T-DXd at 5.4 mg/kg administered as an intravenous (IV) infusion every three-weeks (Q3W) until disease progression, unacceptable toxicity, death, or discontinuation from the study.
  Interventions: Drug: Hydroxychloroquine; Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Hydroxychloroquine — The dosage of hydroxychloroquine is determined based on the dose escalation study, and the appropriate administration method will be determined based on this result.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine Combined With Sacituzumab Govitecan; Hydroxychloroquine Combined With Trastuzumab Deruxtecan
Drug: Sacituzumab Govitecan — Sacituzumab govitecan is a monoclonal antibody, called sacituzumab, linked to a chemotherapy drug, called govitecan. Sacituzumab is a form of targeted therapy because it attaches to specific molecules on the surface of cancer cells, known as Trop-2 receptors, and delivers govitecan to kill them.
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Hydroxychloroquine Combined With Sacituzumab Govitecan; Sacituzumab Govitecan
Drug: Trastuzumab Deruxtecan — Trastuzumab-deruxtecan is a human HER2-directed antibody-drug conjugate (ADC) composed of humanized anti-HER2 immunoglobulin G1 (IgG1) monoclonal antibody (mAb) with the same amino acid sequence as trastuzumab, covalently linked to the membrane-permeable topoisomerase I inhibitor payload, DXd, an exatecan derivative, via a stable tetrapeptide-based linker, selectively cleaved within tumor cells.
  Other Names: DS-8201; Enhertu
  Arms: Hydroxychloroquine Combined With Trastuzumab Deruxtecan; Trastuzumab Deruxtecan

SUMMARY:
Advanced breast cancer is a special subtype of human breast cancer. Conventional guidelines recommend chemotherapy combined with other adjuvant therapies for this subtype of patients. However, the choice of treatment for these patients after treatment progress is a research hotspot in this field. Trastuzumab Deruxtecan (T-DXd) and Sacituzumab Govitecan (SG) are new ADC drugs targeting HER2 or TROP-2 with high efficacy and low toxicity after the progress of first-line treatment. The autophagy agents hydroxychloroquine or chloroquine has become the only FDA (Food and Drug Administration) approved autophagy inhibitor, and hydroxychloroquine and antibody-drug conjugate(ADC) may have synergistic effects based on the previous work results of our research group.

Therefore,we envisage that Trastuzumab Deruxtecan(T-DXd) or Sacituzumab Govitecan (SG) combined with hydroxychloroquine(HCQ) in the treatment of advanced breast cancer in clinical practice has the advantages of improving efficacy and survival.

To this end, we intend to conduct a prospective,multi-center, phase I/II clinical trial to evaluate the efficacy and safety of T-DXd or SG in combination with HCQ in patients with advacned breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent malignant tumor in the world, and 30% of breast cancer patients will enter the advanced stage due to treatment failure. Most patients with advanced breast cancer have had distant organ metastasis, and the median progression free survival period is only 1-2 years.

In the past, advanced breast cancer patients faced the dilemma of poor survival due to the lack of precise targeted therapy. However, through a series of clinical studies, experts in the field of advanced breast cancer have successfully expanded the indications of ADC-based combination targeted therapy from the emergence of first generation ADC to the third generation ADC with "bystander effect", which has significantly prolonged the survival time of patients. Trastuzumab Deruxtecan (T-DXd) and Sacituzumab Govitecan (SG) are new ADC drugs targeting HER2 or TROP-2 with high efficacy and low toxicity after the progress of first-line treatment.

Because both ADC and autophagy involve lysosomes, and the relationship between ADC and autophagy microenvironment has not been elucidated, the combination of autophagy regulators and ADC may be a treatment option that can benefit some patients more.The autophagy agents hydroxychloroquine or chloroquine has become the only FDA (Food and Drug Administration) approved autophagy inhibitor. And the synergistic effect of hydroxychloroquine and antibody-drug conjugate (ADC) has already been confirmed based on preliminary experiments of our research group. We envisage that Trastuzumab Deruxtecan (T-DXd) or Sacituzumab Govitecan (SG) combined with hydroxychloroquine(HCQ) in the treatment of advanced breast cancer in clinical practice has the advantages of improving efficacy and survival.

Therefore, we intend to further validate the efficacy and safety of the Autophagy inhibitor hydroxychloroquine(HCQ) in combination with the latest ADC drugs (T-DXd or SG) in a Phase I/II, randomized, controlled clinical study, in order to provide advanced breast cancer patients with a better choice of precision targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced breast cancer (female, 18 to 70 years old).
2. Pathological confirmed advanced breast cancer.
3. The patient is willing to receive SG or T-DXd treatment.
4. Failure of first-line treatment.
5. Have received no more than 3 chemotherapy schemes for metastatic breast cancer in the past.
6. ECOG physical condition score ≤ 2 points, estimated survival time of no less than 3 months.
7. At least one measurable lesion should be present in the imaging examination within 2 weeks prior to enrollment; Or simple bone metastasis lesions.
8. LVEF≥50%.
9. Previous treatment related toxicity must be relieved to NCI CTCAE (version 5.0) ≤ 1 degree, AST and ALT ≤ 2.5 times the upper limit of normal value, and total bilirubin ≤ 1.5 times the upper limit of normal value.
10. Adequate reserve of bone marrow function: white blood cell count ≥ 3.0 × 10^9/L, neutrophil count ≥ 1.5 × 10^9/L; Platelet count ≥ 100 × 10^9/L; Hemoglobin ≥ 90g/L; Serum creatinine ≤ 1.5 times the upper limit of normal value.

Exclusion Criteria:

1. Patients suffer from various factors such as difficulty swallowing and chronic diarrhea, which affect medication intake and absorption.
2. Individuals with severe heart disease or discomfort, expected inability to tolerate chemotherapy, including but not limited to: fatal arrhythmias or higher-level atrioventricular block, unstable angina, clinically significant valvular heart disease, electrocardiogram showing transmural myocardial infarction, and uncontrolled hypertension.
3. Patients who are known to be allergic to the active ingredients or other components of the investigational drug.
4. Received radiotherapy, chemotherapy, endocrine therapy within 4 weeks prior to enrollment, or is currently participating in any intervention drug clinical trials.
5. Pregnant or lactating women, women of childbearing age who refuse to take effective contraceptive measures during the study period.
6. The researchers believe that patients are not suitable to participate in any other circumstances of this study, which may interfere with the accompanying diseases or conditions of the study, or have any serious medical obstacles that may affect the safety of the subjects.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity, DLT | 3 weeks
  A dose limiting toxicity（DLT）is defined as any of the following-related adverse event(AE) that occurs during the DLT period, graded according to the NCI Common Terminology Criteria for Adverse Events(CTCAE), Version 5.0
Adverse event, AE | 2 years
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Objective Response Rate, ORR | 2 years
  the proportion of patients with a tumor volume reduction of ≥30% and a minimum timeframe according to accepted response evaluation criteria (e.g., RECIST version 1.1 in solid tumors), including cases of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival, PFS | 2 years
  The time from the beginning of treatment to the progression or death of the patient
Overall Survival, OS | 4 years
  The time from the start of randomization to death due to any cause.
Clinical Benefit Rate, CBR | 24 weeks after enrollment
  Proportion of confirmed complete response, partial response, or stable disease ≥ 24 weeks.
Disease Control Rate, DCR | 2 years
  Proportion of patients with stable or shrinking tumor size--sum of the proportions of complete remission (CR), partial remission (PR) and stable disease (SD).
The rate of adverse events | up to 24 weeks after enrollment
  The probability and severity of adverse reactions were analyzed up to 24 weeks after enrollment
Quality of life scale score, QoL | 1 year
  The quality of life score of patients during treatment was analyzed(FACT-B). Performance Status Rating (PSR) was demonstrated for the FACT-B total score, which is the result of the following subscale scores: SWB (the Social / family Well-Being subscale) , EWB (the Emotional Well-Being subscale), AC (Additional Concerns subscale), PWB (the Physical Well-Being subscale), FWB (the Functional Well-Being subscale)
Exploration of biomarkers | the first week after the enrollment
  Objective to explore the correlation between biomarkers and the ORR. The biomarkers will be test by nest-generation sequence, which include 520 genes and tumor mutation burden, like ERBB2/TP53/PIK3CA/ERBB4/CCND1 and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jianli J Zhao, doctorate, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
As personal information of patients is involved, we decided not to share individual participant data of patients.

REFERENCES:
- [Background] Fu Z, Li S, Han S, Shi C, Zhang Y. Antibody drug conjugate: the "biological missile" for targeted cancer therapy. Signal Transduct Target Ther. 2022 Mar 22;7(1):93. doi: 10.1038/s41392-022-00947-7. PMID 35318309
- [Background] Hurvitz SA, Hegg R, Chung WP, Im SA, Jacot W, Ganju V, Chiu JWY, Xu B, Hamilton E, Madhusudan S, Iwata H, Altintas S, Henning JW, Curigliano G, Perez-Garcia JM, Kim SB, Petry V, Huang CS, Li W, Frenel JS, Antolin S, Yeo W, Bianchini G, Loi S, Tsurutani J, Egorov A, Liu Y, Cathcart J, Ashfaque S, Cortes J. Trastuzumab deruxtecan versus trastuzumab emtansine in patients with HER2-positive metastatic breast cancer: updated results from DESTINY-Breast03, a randomised, open-label, phase 3 trial. Lancet. 2023 Jan 14;401(10371):105-117. doi: 10.1016/S0140-6736(22)02420-5. Epub 2022 Dec 7. PMID 36495879
- [Background] Chen YF, Xu YY, Shao ZM, Yu KD. Resistance to antibody-drug conjugates in breast cancer: mechanisms and solutions. Cancer Commun (Lond). 2023 Mar;43(3):297-337. doi: 10.1002/cac2.12387. Epub 2022 Nov 10. PMID 36357174
- [Background] Burris HA 3rd, Rugo HS, Vukelja SJ, Vogel CL, Borson RA, Limentani S, Tan-Chiu E, Krop IE, Michaelson RA, Girish S, Amler L, Zheng M, Chu YW, Klencke B, O'Shaughnessy JA. Phase II study of the antibody drug conjugate trastuzumab-DM1 for the treatment of human epidermal growth factor receptor 2 (HER2)-positive breast cancer after prior HER2-directed therapy. J Clin Oncol. 2011 Feb 1;29(4):398-405. doi: 10.1200/JCO.2010.29.5865. Epub 2010 Dec 20. PMID 21172893
- [Background] Loganzo F, Tan X, Sung M, Jin G, Myers JS, Melamud E, Wang F, Diesl V, Follettie MT, Musto S, Lam MH, Hu W, Charati MB, Khandke K, Kim KS, Cinque M, Lucas J, Graziani E, Maderna A, O'Donnell CJ, Arndt KT, Gerber HP. Tumor cells chronically treated with a trastuzumab-maytansinoid antibody-drug conjugate develop varied resistance mechanisms but respond to alternate treatments. Mol Cancer Ther. 2015 Apr;14(4):952-63. doi: 10.1158/1535-7163.MCT-14-0862. Epub 2015 Feb 2. PMID 25646013
- [Background] Rios-Luci C, Garcia-Alonso S, Diaz-Rodriguez E, Nadal-Serrano M, Arribas J, Ocana A, Pandiella A. Resistance to the Antibody-Drug Conjugate T-DM1 Is Based in a Reduction in Lysosomal Proteolytic Activity. Cancer Res. 2017 Sep 1;77(17):4639-4651. doi: 10.1158/0008-5472.CAN-16-3127. Epub 2017 Jul 7. PMID 28687619
- [Background] Yu SF, Zheng B, Go M, Lau J, Spencer S, Raab H, Soriano R, Jhunjhunwala S, Cohen R, Caruso M, Polakis P, Flygare J, Polson AG. A Novel Anti-CD22 Anthracycline-Based Antibody-Drug Conjugate (ADC) That Overcomes Resistance to Auristatin-Based ADCs. Clin Cancer Res. 2015 Jul 15;21(14):3298-306. doi: 10.1158/1078-0432.CCR-14-2035. Epub 2015 Apr 3. PMID 25840969
- [Background] Le Joncour V, Martins A, Puhka M, Isola J, Salmikangas M, Laakkonen P, Joensuu H, Barok M. A Novel Anti-HER2 Antibody-Drug Conjugate XMT-1522 for HER2-Positive Breast and Gastric Cancers Resistant to Trastuzumab Emtansine. Mol Cancer Ther. 2019 Oct;18(10):1721-1730. doi: 10.1158/1535-7163.MCT-19-0207. Epub 2019 Jul 10. PMID 31292166
- [Background] Li X, He S, Ma B. Autophagy and autophagy-related proteins in cancer. Mol Cancer. 2020 Jan 22;19(1):12. doi: 10.1186/s12943-020-1138-4. PMID 31969156
- [Background] Mauthe M, Orhon I, Rocchi C, Zhou X, Luhr M, Hijlkema KJ, Coppes RP, Engedal N, Mari M, Reggiori F. Chloroquine inhibits autophagic flux by decreasing autophagosome-lysosome fusion. Autophagy. 2018;14(8):1435-1455. doi: 10.1080/15548627.2018.1474314. Epub 2018 Jul 20. PMID 29940786
- [Background] Yamamoto K, Venida A, Yano J, Biancur DE, Kakiuchi M, Gupta S, Sohn ASW, Mukhopadhyay S, Lin EY, Parker SJ, Banh RS, Paulo JA, Wen KW, Debnath J, Kim GE, Mancias JD, Fearon DT, Perera RM, Kimmelman AC. Autophagy promotes immune evasion of pancreatic cancer by degrading MHC-I. Nature. 2020 May;581(7806):100-105. doi: 10.1038/s41586-020-2229-5. Epub 2020 Apr 22. PMID 32376951